CLINICAL TRIAL: NCT01600261
Title: iCam Clinical Validation Study
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-47425
Record Dates: First submitted 2012-05-14; First posted 2012-05-17 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Eye Disease
Keywords: without eye disease
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- eye exam

SUMMARY:
Comparison study to assess photo image quality of a new color fundus camera compared to that of a commercially available color fundus camera.

DETAILED DESCRIPTION:
Optovue has developed a new color fundus camera for imaging the eye with up to 45 degree field of view and without the use of dilating drops. The purpose of the study is to compare the image quality of the new camera with that of a commercially available color fundus camera. Consented subjects will undergo a general ophthalmic examination and series of fundus photography exams using the study device and comparison device. Photo image quality will be assessed for determination of clinically usefulness.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able and willing to complete the required examination

Exclusion Criteria:

* Spherical Equivalent outside -12 diopter to +15 diopter
* Without lens
* Inability to fixate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects shall be recruited from the practice of the principal investigator (PI).
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
proportion of clinically useful images | Day 1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Livermore Optometry Group, Livermore, California
  - Buena Vista Eye Care, San Jose, California